CLINICAL TRIAL: NCT02945137
Title: Comparison of Rapid Urease Test Between the Gastric Body and Antrum in Helicobacter Pylori-Infected Stomach
Brief Title: Optimal Site for Rapid Urease Test in the Stomach
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Assistant Professor, Soonchunhyang University Hospital
Other Study IDs: SCHDDC 2016-10
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biospecimen would be obtained for urease test (commercial name: CLOtest).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The accurate diagnosis of H. pylori infection is an important step for establishing the strategy for gastric cancer prevention. During endoscopy, rapid urease test (RUT) is the first of biopsy-based H. pylori tests. Despite indirect test for H. pylori detection, RUT shows rapid result with good sensitivity and specificity. Several study reported that H. pylori density was related to positive reaction time of RUT. However, there was no study comparing the positive reaction times of RUT according to biopsy site, degree of gastric atrophy, and intestinal metaplasia.

DETAILED DESCRIPTION:
The aims of this study were to: (1) assess the positive reaction times of RUT in the body and antrum, (2) investigate the association between the difference of RUT results (body and antrum) and gastric atrophy, and intestinal metaplasia, and (3) evaluate the optimal biopsy site for RUT according to degree of gastric atrophy in Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent upper endoscopy and rapid urease test

Exclusion Criteria:

* : age < 20 or > 70 years; anemia (serum hemoglobin level < 10 g/dL); severe systemic disease or advanced chronic liver disease; use of certain medications, including proton pump inhibitors, H2-receptor antagonists, or antibiotics; a history of H. pylori eradication; a history of gastric surgery; a recent history of upper gastrointestinal bleeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects who underwent an upper gastrointestinal endoscopy were enrolled in this study at a single, tertiary-care, academic medical center. During endoscopy, rapid urease tests would be performed in the body and antrum.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Positive reaction time of urease test | within 24 hours
  Color change to red or pink means positivity

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Assistant Professor
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No